CLINICAL TRIAL: NCT01344109
Title: A Pilot Study of Tumor-Derived Exosomes as Diagnostic and Prognostic Markers in Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Withdrawn | Type: Observational
Why Stopped: Lab company that was to do testing was sold
Sponsor: Leo W. Jenkins Cancer Center (Other)
Responsible Party: Principal Investigator, Susan E. Eubanks, RN, MSN, OCN, Clinical Trials Manager, Leo W. Jenkins Cancer Center
Other Study IDs: ECU 003
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum will be centrifuged to plasma which will be transferred to alliquots, and frozen prior to shipping. Exosomes will be extracted from the frozen plasma with half of the sample used for antibody testing and the remaining sample will be used for RNA analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast cancer patients: Newly diagnosed patients with breast cancer presenting with operable breast tumor prior to initiation of of neoadjuvant chemotherapy (choice of chemotherapy will be the the treating physician's discretion)
- Healthy volunteers: Adult women without a cancer diagnosis.

SUMMARY:
This is a pilot study evaluating the use of tumor derived exosomes as a marker for response to therapy in women receiving neoadjuvant chemotherapy for newly diagnosed breast cancer. Tumor derived exosome analysis may be a novel diagnostic and prognostic biosignature in breast cancer, which could prove to be a tool for earlier diagnosis, more effective treatments, and improved markers of response in order to increase survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Women with biopsy proven invasive carcinoma of the breast
* Women with locally advanced breast cancer and breast tumors measuring >/= 2cm who are deemed candidates for preoperative chemotherapy
* Age >/= 18 years old
* Expected survival >/= 6 months
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2 at initiation of study
* Initial required laboratory values:

Absolute neutrophil count >/= 1.5 x 10(9)/L Platelet count >/= 100,000 x 10(9)/L Creatinine clearance >/= 50mL/min (calculated by Cockcroft-Gault method) Liver function tests (AST, ALT, total bilirubin) </= 2.5 x ULN Urine or serum HCG negative (if female of childbearing potential)

* Women may be enrolled on ongoing therapeutic preoperative chemotherapy trials

Exclusion Criteria:

* No prior chemotherapy for breast cancer
* No limitations for prior radiation therapy
* No active, serious infection or medical or psychiatric illness likely to interfere with participation in this trial
* Non-pregnant and non-nursing patients only. Patients of reproductive potential must agree to use an effective means of birth control
* No prior liver transplant or bone marrow transplant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed breast cancer patients prior to neoadjuvant chemotherapy treatment and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To characterize protein surface markers and RNA profiles in tumor derived exosomes from breast cancer patients undergoing neoadjuvant chemotherapy | up to 2 years from start of study
  Compare tumor derived exosomes at baseline, monthly during chemotherapy, at the completion of chemotherapy treatment, and after surgery to determine residual cancer burden. Tumor derived exosome expression will be correlated with both clinical and pathologic response.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Raab, MD, Principal Investigator — Brody School of Medicine at ECU
Locations (1):
- Leo W. Jenkins Cancer Center, Greenville, North Carolina, United States